CLINICAL TRIAL: NCT03286010
Title: Cluster Randomization Trial of Peer Support for Women With Heart Disease: Women@ Heart
Brief Title: Peer Support for Women With Heart Disease: Women@Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170613-01H
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Coronary Heart Disease; Women's Health
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the W@H group will be assembled in small groups of 6-12 participants and attend 12-biweekly sessions over a 24-week intervention period. The sessions will be led by a trained peer leader and will be held in a variety of convenient locations in close geographic proximity to participants' home postal codes. Participants will receive a manual containing copies of learning exercises and educational material. Session content is focused on: emotional support (sharing your story, road to recovery, exploration of feelings, coping with changes, emotional management, coping with distress, effective communication, empowerment); informational support (self care behaviours, risk factor education and management, health care system and community resource navigation); and appraisal support (goal setting, action planning, problem solving, relapse prevention).
  Interventions: Behavioral: Women@Heart Program
- Control (No Intervention): Participants in the control group will be eligible to participate in the study, but cannot participate because there are no groups within their geographical region. They will be offered the W@H program after their 26-week follow up.

INTERVENTIONS:
Behavioral: Women@Heart Program — The Women@Heart program is taught by trained peer leaders. Session content is focused on: emotional support (sharing your story, road to recovery, exploration of feelings, coping with changes, emotional management, coping with distress, effective communication, empowerment); informational support (self care behaviours, risk factor education and management, health care system and community resource navigation); and appraisal support (goal setting, action planning, problem solving, relapse prevention). In total there are 12-biweekly sessions offered over a 24-week period.
  Arms: Intervention

SUMMARY:
Women with heart disease are more likely to die or suffer another cardiac event or stroke within 5 years of an index event compared to men. They are also more likely to suffer depression and report lower quality of life. Cardiac Rehabilitation programs have been designed to address these issues, but most women do not attend. Women indicate they have a greater need to talk about their experiences with heart disease and seek social support to help them cope. Peer support, the assistance provided by other women with a similar illness experience, may be one way to enhance social support for women with heart disease and help them improve their psychosocial well-being. The Investigators have developed a peer support program called Women@Heart (W@H). The program is led by trained peer leaders (women who themselves have made a successful recovery from a heart event). A pilot test of the program showed promising results. The Investigators now need to conduct a more rigorous evaluation of the program.

The main objective of this project is to determine if the W@H program helps women to improve their psychosocial well-being compared to being on a waiting list to participate in the program. It will also examine the effect of the program on: health behaviours (tobacco smoking, physical activity, sedentary behaviour, fruit and vegetable consumption, and medication adherence); coronary risk factors; and clinical outcomes (re-hospitalization, health care system use, death).

ELIGIBILITY:
Inclusion Criteria:

1. Women who have been hospitalized at UOHI in the past year with stable CHD, including: AMI; stable angina with corroborating evidence of CHD; recent CABG; or percutaneous coronary intervention (to allow examination of mechanisms linking the intervention and psychosocial well-being with health and healthcare outcomes);
2. Women ≥ 18 years of age (the age of consent in Ontario);
3. Women able to read and understand English or French;
4. Women who reside in Ontario and are eligible for Ontario Health Insurance Plan (to permit linkage with administrative data housed at the Institute for Clinical Evaluative Sciences [ICES]);
5. Women available to participate over the next 6 months (the intervention and data collection takes place over this time frame -- reducing the probability of missing data);
6. Women able to provide informed consent.

Exclusion Criteria:

1. Women who have been hospitalized primarily for valve replacement or repair, HF, pulmonary hypertension, endocarditis or pericarditis (to reduce heterogeneity and avoid confounding when examining mechanisms linking the intervention and psychosocial well-being with health and healthcare outcomes);
2. Women who, in the opinion of the UOHI clinical psychologist, manifest psychiatric illness or cognitive impairment that would preclude participation in W@H (i.e. they are unable to benefit from the intervention, to prevent disruption of other participants).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Psychosocial well-being as measured by a total composite score | Baseline to week 26 follow up
  The composite score will combine data from seven measures (ESSI, BCI, BAI, BDI2, MCS, HeartQol and PSS)

SECONDARY OUTCOMES:
Smoking Status | Baseline to week 26 follow up
  Measured by self report and carbon monoxide breath test
Fruit/Vegetable consumption | Baseline to week 26 follow up
  Measured by two questions from the Ontario Health Study that assess typical daily servings of fruits and vegetables.
Menstrual Status | Baseline to week 26 follow up
  Measured through self reported menstrual status (i.e., pre, peri or post-menopausal)
Gender Role Identity | Baseline to week 26 follow up
  The BEM Sex Role Inventory will be used to assess participants' feelings towards their own gender role identities (masculine, feminine, androgynous and undifferentiated).
Physical Activity | Baseline to week 26 follow up
  Measured through self reported physical activity
Salt Consumption | Baseline to week 26 follow up
  Assessed using 1 question from the Canadian Community Health Survey (2015) that assess weekly intake of salty foods.
Medication Adherence | Baseline to week 26 follow up
  Assessed through two questions asking whether or not participants ever forget to take their medication and if they ever stop taking their medication (if so why).

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Mullen, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No